CLINICAL TRIAL: NCT03358160
Title: Motor Representations in Orthopedic Patients: Pilot Studies
Brief Title: Motor Representations in Orthopedic Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: RMPO
Record Dates: First submitted 2017-11-21; First posted 2017-11-30 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Orthopedic Disorder; Motor Disorder; Perceptual Disorders
MeSH Terms: conditions — Musculoskeletal Diseases; Motor Disorders; Perceptual Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- TKA: Orthopaedic patients who underwent surgical operation for total knee arthroprothesis.
  Interventions: Behavioral: Action discrimination tasks.
- Rizoarthrosis: Orthopaedic patients who underwent surgical operation to treat chronic arthrosis of the thumb.
  Interventions: Behavioral: Action discrimination tasks.
- Healthy Controls: Healthy age-matched controls.
  Interventions: Behavioral: Action discrimination tasks.

INTERVENTIONS:
Behavioral: Action discrimination tasks. — The investigators will compare the groups' performance during action discrimination tasks related to movements of the upper vs. lower limbs.

SUMMARY:
The aim of this study is to investigate the possible effects that a motor limitation at the peripheral level might have on the ability to visually discriminate others' actions.

Previous literature has shown that specific motor skills (motor expertise) facilitate the visual discrimination of domain-specific actions, and that these motor experts' superior abilities might be mediated by areas not only responsible for the visual recognition of movements (as it happens in non-expert subjects) but also involved in motor planning. Similarly, impairment in the motor system due to neurological damage modulates not only the ability to perform movements but also the ability to discriminate and predict the temporal course of observed actions.

Based on these findings, it has been hypothesized that the motor representations of gait, despite being a hyper-learned motor pattern, might be subjected to modification as a result of an impairment of walking caused by a peripheral functional limitation in the lower limbs as the one characterizing orthopaedic patients who underwent a surgical operation for total knee arthroprosthesis. In this protocol, patients are thus required to perform visual discrimination tasks based on the observation of movements performed with either the upper or lower limbs, and their performance is expected to correlated with their functional impairments in movement execution.

These results would indicate that the (in)ability to perform a movement might have an impact on its representation at the central level and on internal motion simulation capabilities, which also influence the ability to visual discriminate others' actions through action-perception transfer: this would suggest that rehabilitation in orthopaedic patients should take into account (and restore) such a central impairment in motor representations.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be able to understand instructions and have no history of neurological or psychiatric disorders.

Exclusion Criteria:

* History of neurological or psychiatric disorders.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Orthopaedic patients and age-matched healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-05-31 (Actual); Primary Completion 2017-03-30 (Actual); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Group Differences in action discrimination performance. | End 2018.
  Group Differences in action discrimination performance depending on the impairment in movement execution.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Galeazzi Orthopedic Hospital, Milan, Italy